CLINICAL TRIAL: NCT05240222
Title: A Theory-Informed Pre-Implementation Enhancement Strategy Targeting Mechanisms and Outcomes of Implementation: A Triple-Blind Randomized Controlled Trial
Brief Title: Pre-Implementation Enhancement Strategy To Improve Teachers' Intention to Implement Evidence-Based Practices
Acronym: SC-PIES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: University of Washington (Other); University of Minnesota (Other)
Responsible Party: Principal Investigator, Yanchen Zhang, Assistant Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: PIES001
Record Dates: First submitted 2022-01-10; First posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Child Behavior Disorders; Implementation Science; Adolescent Problem Behavior at School; Healthcare Providers
Keywords: Implementation Science; School Mental Health Services; Healthcare Providers; School Teachers
MeSH Terms: conditions — Child Behavior Disorders

STUDY DESIGN:
Intervention Model Description: This is a triple-blind parallel randomized controlled trial. Specifically, teachers from a diverse urban district were recruited and randomly assigned to either the treatment (SC-PIES) or active control condition (administrative meeting). Based on the condition assigned, teachers received the SC-PIES (or met with administrators) before EBP training. The investigators assessed teachers' ITI, intervention fidelity, and youth behavioral outcome (academic engagement as an incompatible behavior to externalizing disorders) before treatment, immediately after training, and six weeks afterward.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All personnel involved in this study were masked, including the participating teachers, investigators, trainers who deliver the SC-PIES or meeting, and staff who collected the outcome data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Theory-informed pre-implementation enhancement strategies (SC-PIES) (Experimental): The SC-PIES was delivered to teachers as a one-hour professional development session immediately before receiving specific training about evidence-based student behavioral management practices and subsequent follow-up consultation. The content of SC-PIES was grounded in three social-cognitive principles: (a) growth mindset, (b) saying-is-believing, and (c) commitment and consistency.
  Interventions: Behavioral: Pre-implementation enhancement strategies (SC-PIES)
- Active control (Sham Comparator): Participants in the active control condition will meet with school administrators to talk about their work irrelevant to SC-PIES or student behaviors. The meeting lasted for the same duration as the SC-PIES at the same time as those in the treatment condition.
  Interventions: Other: Sham comparator

INTERVENTIONS:
Behavioral: Pre-implementation enhancement strategies (SC-PIES) — The SC-PIES was delivered to teachers as a one-hour professional development session immediately before receiving specific training about evidence-based student behavioral management practices and follow-up consultation. SC-PIES content was grounded in three social-cognitive principles: (a) growth mindset, (b) saying-is-believing, and (c) commitment and consistency.
  Arms: Theory-informed pre-implementation enhancement strategies (SC-PIES)
Other: Sham comparator — Participants in the active control condition will meet with school administrators to talk about their work irrelevant to SC-PIES or student behaviors. The meeting lasted for the same duration as the SC-PIES at the same time as those in the treatment condition.
  Arms: Active control

SUMMARY:
Background: As the most common setting where youth access behavioral health services, the education sector frequently employs training and follow-up consultation as cornerstone implementation strategies to promote the uptake and use of evidence-based practices (EBPs), which are often insufficient to produce desired implementation outcomes (e.g., intervention fidelity) and changes in youth behavioral health outcomes (e.g., reduced externalizing behaviors). There is a need for theoretically-informed pre-implementation enhancement strategies (PIES) that increase the yield of training and follow-up consultation. Specifically, social-cognitive theory explicates principles to inform the design of strategy content and specific mechanisms of behavior change, such as intentions to implement (ITI), to target via a PIES that increase provider to more active implementation strategies. Methods: This triple-blind randomized controlled trial preliminarily examined the efficacy of a pragmatic PIES (SC-PIES) to improve the implementation of universal EBPs in the education sector. Participants were randomly assigned to the treatment (PIES) or active control condition (meeting with administrators). The investigators assessed participants' ITI, intervention fidelity, and youth behavioral health outcome before, immediately after, and six-week following treatment.

DETAILED DESCRIPTION:
1. Background and study aims:

   As the most common setting where youth access behavioral health services, the education sector frequently employs training and follow-up consultation as cornerstone implementation strategies to promote the uptake and use of evidence-based practices (EBPs). However, these strategies alone are not sufficient to promote the desired implementation (e.g., intervention fidelity) and youth behavioral health outcomes (e.g., externalizing behaviors). Theory-informed pragmatic pre-implementation enhancement strategies (PIES) are needed to increase the yield of training and consultation. Specifically, social-cognitive theory explicates principles to inform the design of strategy content and specific mechanisms of behavior change (e.g., "intentions to implement"; ITI) to target to increase providers' responsiveness to training and consultation. This triple-blind parallel randomized controlled trial preliminarily examined the efficacy of a pragmatic PIES based on social-cognitive theories (SC-PIES) to improve the implementation and youth outcomes of universal EBPs in schools. Four aims will be examined:
   1. As compared to control, does the pre-implementation enhancement strategy based on social-cognitive theories (SC-PIES) significantly improve teachers' implementation intentions to implement PCBM practices at posttest after adjusting baseline and covariates?
   2. As compared to control, is receiving SC-PIES associated with significantly improved teachers' intervention fidelity and class-wide youth behavioral health outcome at the 6-week follow-up after adjusting for baseline and covariates?
   3. Does teachers' intention to implement mediate the association between study condition and intervention fidelity?
   4. Does teachers' intervention fidelity mediate the association between their intentions to implement and class-wide youth behavioral health outcomes?
2. Who can participate? Any teacher who has no prior training about or experience of implementing Proactive Classroom Behavioral Management Strategies (PCBM) targeting youth behaviors in a school district. No restriction on age, gender, experience, or other demographic variables.
3. What does the study involve? The participating teachers will be randomly assigned to either the treatment (SC-PIES) or active control condition (administrative meeting). The SC-PIES was delivered to teachers as a one-hour professional development session immediately before receiving specific training about evidence-based PCBM practices and subsequent follow-up consultation. Teachers in the active control condition will meet with their administrators to talk about their work irrelevant to SC-PIES or student behaviors. The investigators assessed teachers' ITI, intervention fidelity, and youth behavioral outcome (academic engagement as an incompatible behavior to externalizing disorders) before treatment, immediately after training, and six weeks afterward.
4. What are the possible benefits and risks of participating? Teachers participating in this study will benefit from expert training and consultation to improve their intentions and skills to implement a set of EBPs to help their students' behavioral problems. No risks to participants were expected based on relevant literature in education and implementation science.

ELIGIBILITY:
Inclusion Criteria:

* Teachers who have no prior training about Proactive Classroom Behavioral Management Strategies (PCBM) targeting youth behaviors in an urban school district.
* Teachers who have no prior experience in implementing Proactive Classroom Behavioral Management Strategies (PCBM) targeting youth behaviors in an urban school district.

Exclusion Criteria:

* Teachers who have attended more than three training sessions about Proactive Classroom Behavioral Management Strategies (PCBM) targeting youth behaviors in an urban school district.
* Teachers who have more than one month of experience in implementing Proactive Classroom Behavioral Management Strategies (PCBM) targeting youth behaviors in an urban school district.

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-07-22 (Actual); Primary Completion 2017-05-20 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Teachers' Intentions to Implement (ITI) at 3 Days | Three days following the baseline test of teachers' intentions to implement
  The Modified Intentions to Use Scale was adopted to assess the change in teachers' intentions to implement from baseline to immediate post-test. The scale is originally developed from research on practitioners' intention to adhere to measurement-based care and is consistent with the recommendations for assessing behavioral intentions based on the theory of planned behavior (Godin & Kok, 1996). The scale consists of five items on a 7-point Likert scale ranging from "greatly disagree" to "greatly agree". The items were modified to specifically assess teachers' intentions to implement EBPs. The scale showed acceptable reliability and validity in prior research.
Change from Baseline Teachers' Intervention Fidelity at 6 weeks. | Six weeks following the baseline test of teachers' intervention fidelity
  A team of trained professionals, who were blinded to the random assignment results, conducted structured observations to assess the intervention fidelity, which is operationalized in this study as "adherence to core components of the classroom management practices". The data collection took place at pre-test and 6-week follow-up to allow enough time to detect and compare changes in intervention fidelity. First, during core instructional times, trained observers observed two occasions at pre-test and 6-week follow-up to code the presence or absence of the core components of the evidence-based practices. Immediately following the observations, these observers completed a fidelity rating rubric, which was created by operationalizing three core components of each PCBMs such that observers could reliably observe and rate them. The average of the observation coding and the rubric scores represents each teacher's fidelity.

SECONDARY OUTCOMES:
Change from Baseline Students' Academic Engaged Time (AET) at 6 weeks | Six weeks following the baseline test of students' AET
  AET is defined as "any instance where youths are attending to instruction, watching the teacher or speaker, or concentrating on their classwork". This study will use Direct Behavior Ratings (DBRs) for academic engaged time (AET) with which a teacher observes a youth's AET throughout a predetermined interval. Based on the literature of DBRs, teacher-completed DBRs have strong correlations to Structured Direct Observation in assessing AET (Sanetti, 2009). The DBRs will be completed at pre-test and 6-week follow-up. For comparability across classrooms, each teacher completes DBRs during the reading/language arts block at the same time each day of the week for five randomly selected youths, whose results will be then averaged for that class. This approach has demonstrated adequate reliability and validity to capture class-wide AET in education literature (Sanetti, 2009).

CONTACTS AND LOCATIONS:
Overall Officials: Yanchen Zhang, PhD, Principal Investigator — University of Iowa

IPD SHARING:
Plan to Share IPD: Yes
The de-identified datasets generated and analyzed during the current study are available in the Open Science Framework repository, [osf.io/d5t4m/].
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: From December 1st, 2021 with no ending date
Access Criteria: Public upon request to the principle investigator
URL: http://osf.io/d5t4m/

REFERENCES:
- [Background] Godin G, Kok G. The theory of planned behavior: a review of its applications to health-related behaviors. Am J Health Promot. 1996 Nov-Dec;11(2):87-98. doi: 10.4278/0890-1171-11.2.87. PMID 10163601
- [Background] Sanetti LM, Kratochwill TR. Toward developing a science of treatment integrity: Introduction to the special series. School Psychology Review. 2009 Dec 1;38(4):445.
- [Derived] Zhang Y, Cook CR, Azad GF, Larson M, Merle JL, Thayer J, Pauls A, Lyon AR. A Pre-Implementation Enhancement Strategy to Increase the Yield of Training and Consultation for School-Based Behavioral Preventive Practices: a Triple-Blind Randomized Controlled Trial. Prev Sci. 2023 Apr;24(3):552-566. doi: 10.1007/s11121-022-01464-3. Epub 2022 Nov 11. PMID 36367633
- Available data/document: Individual Participant Data Set: DOI 10.17605/OSF.IO/D5T4M — http://osf.io/d5t4m/ — The de-identified datasets generated and analyzed during the current study are made available in the Open Science Framework repository, [osf.io/d5t4m/].